CLINICAL TRIAL: NCT04699019
Title: Evaluating the Foot Touch Framework Model in Running
Brief Title: Evaluating the Foot Touch Framework Model
Status: Completed | Type: Observational
Sponsor: Orthocare Innovations, LLC (Industry)
Collaborators: FastEquation Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20190314
Record Dates: First submitted 2020-12-22; First posted 2021-01-07 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Barefoot Running

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active Runners: All participants will be required to run unshod for a combination of four prescribed speeds (walking and up to 9 mph) and three different foot strike patterns (rearfoot, midfoot, and forefoot) on level ground.
  Interventions: Other: Four speeds; Other: Foot Strike Pattern

INTERVENTIONS:
Other: Four speeds — Four speeds ranging from a set walking speed up to 9 mph
Other: Foot Strike Pattern — Foot strike sequences (rearfoot strike, midfoot strike, forefoot strike)

SUMMARY:
A Foot Touch framework model has been developed to express the ground reaction force waveforms observed for walking and running. The purpose of this research is to collect ground reaction force data during walking and running that can be used to evaluate and verify the Foot Touch framework.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women
* Capable of independently walking and running at various speeds for a minimum of 30 minutes
* No history of significant injuries in the past six months
* Ability to walk and run without shoes/footwear
* Ability to perform one- and two-footed hops up and down from 5 cm and 10 cm heights
* Ability to provide informed consent

Exclusion Criteria:

* Confounding chronic injury or musculoskeletal problem
* Pregnancy
* Symptomatic cardiovascular disease or chronic obstructive pulmonary disease
* Not able to read and understand English

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, able-bodied participants will be recruited from the general public.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-07-28 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
MatScan Forces | Assessed on day 1 (data collection day)
  Ground reaction forces for distinct anatomical regions of the foot (Calcaneal, Tarsal, Metatarsal, Phalangeal) measured by the MatScan system

SECONDARY OUTCOMES:
Ground reaction force | Assessed on day 1 (data collection day)
  Ground reaction force measured by the force plate during walking, running, and hopping tasks
Ankle joint angle | Assessed on day 1 (data collection day)
  Ankle joint angle measured by motion analysis system during walking, running, and hopping tasks
Knee joint angle | Assessed on day 1 (data collection day)
  Knee joint angle measured by motion analysis system during walking, running, and hopping tasks
Hip joint angle | Assessed on day 1 (data collection day)
  Hip joint angle measured by motion analysis system during walking, running, and hopping tasks

CONTACTS AND LOCATIONS:
Locations (1):
- Orthocare Innovations, LLC, Edmonds, Washington, United States

IPD SHARING:
Plan to Share IPD: No